CLINICAL TRIAL: NCT05082389
Title: Prediction of Hospital Readmissions in SAPV (Specialised Home Palliative Care) Patients - Identification of Structural Factors and Support Needs of Family Caregivers
Brief Title: Prediction of Hospital Readmissions in SAPV (Specialised Home Palliative Care) Patients
Acronym: PRePP
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: University Hospital Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: BO-EK-320072020
Record Dates: First submitted 2021-05-04; First posted 2021-10-19 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Palliative Care
Keywords: Patient reported outcome (PRO); family caregivers; specialized palliative home-based care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Specialised outpatient palliative care (German: Spezialisierte ambulante Palliativversorgung, abbreviation: SAPV) aims to support incurably ill or dying people spending their last lifetime at home. Furthermore, a major goal is to prevent unnecessary hospital admissions. However, they occasionally occur for various reasons. This project aims to explore predictors of readmission in terms of structural factors as well as family caregivers' psychological distress.

Study Aims

1. Identification of structural predictors and caregiver reported predictors for hospital readmissions.
2. Identification of psychological liabilities of nursing relatives.
3. Developing a concept to support nursing relatives.

DETAILED DESCRIPTION:
1. Background Specialised outpatient palliative care (German: Spezialisierte ambulante Palliativversorgung, abbreviation: SAPV) aims to support incurably ill or dying people spending their last lifetime at home if possible.

   At the same time unnecessary hospital readmissions should be prevented. However, they occasionally occur for various reasons. Due to an analysis of own data including 81 patient of our institution we found the following structural factors influencing hospital readmissions: On average there are 1.3 hospital admissions per patient while receiving palliative care. The quality of home-based care is one factor for hospital readmission. Especially patients´ high symptom burden as well as caregivers´ report of depression and anxiety lead to unplanned hospital readmissions.

   Former studies show a major impact of psychosocial pressure of relatives, for example sadness, sorrows, and exhaustion). High scores of distresses seem to correlate with a higher number of unfulfilled needs. About one third of the nursing relatives reached high scores concerning anxiety and depression. Moreover, an elevated level of resilience relates to a positive opinion of health, better social support, and a decreased rate of depressions of patients who suffer from metastasised oncological diseases. Life quality of nursing relatives is not only decreased in a psychological way but in all parts of life and is influenced by spiritual well-being and by the relation of the patient and the nursing person. The relevance of stable relationship between familiar and professional helpers is also described by Roen and his colleagues.
2. Methods This study is designed as a single-arm, single institution, non-randomized observational study.

The primary study aim is to investigate structural, and caregiver reported reasons for hospital readmission. Burden and needs for support of informal caregivers that lead to a failure of ambulatory care should be identified. Afterwards experts will develop strategies to improve the identified factors and therefore reduce the number of unnecessary hospital readmissions.

2.1 Primary goal Are there any structural or caregiver reported factors influencing hospital readmission during concomitant care by SAPV?

2.2 Secondary goals To explore the burden and supportive-care needs experience informal caregivers caring for patients with an incurable and progressive disease at home? Which concepts can be developed to improve pressures and needs for support of nonprofessional caregivers during the patients´ palliative care?

2.3 Patients This study aims to include consecutively 240 patients of our institution's specialized outpatient palliative care team.

2.4 Primary and Secondary endpoints Primary outcome is the number of unplanned admissions. An unplanned admission is defined as any hospital stay not being previously planned as part of intended treatment.

Secondary endpoints include structural data taken from the patients´ medical records. Furthermore, four validated questionnaires will be administered to obtain family caregiver reported factors:

* quality of life (WHOQOL BREF (WHO | WHO Quality of Life-BREF (WHOQOL-BREF), n.d.)
* psychological distress (NCCN Distress Thermometer)
* anxiety (Generalized Anxiety Disorder 7-item scale)
* depression (Health Questionnaire depression module 9- item scale).

In addition, a non-standardized questionnaire identifying the burden of relatives caused by the SARS-CoV-2-pandemia is administered.

The following structural data concerning the informal caregiver will be evaluated: age, sex, relationship to the patient, amount of care, educational background, and actual working situation.

The following structural data concerning the patient will be registered: age, sex, diagnosis justifying imbursement of palliative care, duration of palliative care, hospital admissions during SAPV, support by informal caregivers, level of care, use of home-based services, home hospice, reason for hospital admissions, concomitant cancer therapy, data concerning the hospital admission, place of discharge. Information will be collected from the patients´ medical records.

Nurses of SAPV will answer surprise questions monthly: There will be one surprise question concerning patients´ death and another one concerning the probability of hospital readmission.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (>17years)
* with advanced, non-curable disease with limited life expectancy and complex symptoms
* treated by a Specialised Home Palliative Care - team
* providing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients treated in SAPV University hospital Dresden will be investigated by descriptive statistics. All respective non-professional-caregivers will be asked to take part in the survey. They must meet the aforementioned inclusion criteria and provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Circumstances of Unplanned hospital admission | 18 months
  Hospital admission not intended and/or planned by either professional nor non-professional care givers

SECONDARY OUTCOMES:
Quality of Life of primary non-professional care-giver | 18 months
  Quality of Life as assessed by WHOQOL-BREF (World Health Organization Quality of Life)
Psychological Distress of primary non-professional care-giver | 18 months
  Psychological Distress as assessed by NCCN-Distress Thermometer
Anxiety of primary non-professional care-giver | 18 months
  Anxiety as assessed by the Generalized Anxiety Disorder 7-item scale
Depressivity of primary non-professional care-giver | 18 months
  Depressivity as assessed by the Health Questionnaire depression module 9-item scale
Characteristics of the non-professional care-giver | 18 months
  Characteristics of primary non-professional care giver such as age, gender, kind of relation to the patient, duration of daily care, highest education, employment status
Characteristics of patient | 18 months
  Characteristics of patient such as age, gender, diagnosis, duration of previous hospitalisation, additional supportive services, number of visits by SAPV, symptoms status,

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Schütte, MD, Principal Investigator — University Hospital Dresden; Palliative Care Unit; Leopold Hentschel, Dipl.-Psych., Principal Investigator — University Hospital Dresden; Department of Psychooncology
Locations (1):
- University Hospital Carl Gustav Carus, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ullrich A, Ascherfeld L, Marx G, Bokemeyer C, Bergelt C, Oechsle K. Quality of life, psychological burden, needs, and satisfaction during specialized inpatient palliative care in family caregivers of advanced cancer patients. BMC Palliat Care. 2017 May 10;16(1):31. doi: 10.1186/s12904-017-0206-z. PMID 28486962
- [Background] Gotze H, Brahler E, Gansera L, Schnabel A, Gottschalk-Fleischer A, Kohler N. Anxiety, depression and quality of life in family caregivers of palliative cancer patients during home care and after the patient's death. Eur J Cancer Care (Engl). 2018 Mar;27(2):e12606. doi: 10.1111/ecc.12606. Epub 2016 Nov 17. PMID 27859889
- [Background] Halkett GKB, Lobb EA, Shaw T, Sinclair MM, Miller L, Hovey E, Nowak AK. Do carer's levels of unmet needs change over time when caring for patients diagnosed with high-grade glioma and how are these needs correlated with distress? Support Care Cancer. 2018 Jan;26(1):275-286. doi: 10.1007/s00520-017-3846-x. Epub 2017 Aug 14. PMID 28808797
- [Background] Hwang IC, Kim YS, Lee YJ, Choi YS, Hwang SW, Kim HM, Koh SJ. Factors Associated With Caregivers' Resilience in a Terminal Cancer Care Setting. Am J Hosp Palliat Care. 2018 Apr;35(4):677-683. doi: 10.1177/1049909117741110. Epub 2017 Nov 15. PMID 29141459
- [Background] Spatuzzi R, Giulietti MV, Ricciuti M, Merico F, Fabbietti P, Raucci L, Bilancia D, Cormio C, Vespa A. Exploring the associations between spiritual well-being, burden, and quality of life in family caregivers of cancer patients. Palliat Support Care. 2019 Jun;17(3):294-299. doi: 10.1017/S1478951518000160. Epub 2018 May 11. PMID 29749317
- [Background] Kobayakawa M, Ogawa A, Konno M, Kurata A, Hamano J, Morita T, Kizawa Y, Tsuneto S, Shima Y, Aoyama M, Miyashita M. Psychological and psychiatric symptoms of terminally ill patients with cancer and their family caregivers in the home-care setting: A nation-wide survey from the perspective of bereaved family members in Japan. J Psychosom Res. 2017 Dec;103:127-132. doi: 10.1016/j.jpsychores.2017.10.012. Epub 2017 Oct 23. PMID 29167039
- [Background] Roen I, Stifoss-Hanssen H, Grande G, Brenne AT, Kaasa S, Sand K, Knudsen AK. Resilience for family carers of advanced cancer patients-how can health care providers contribute? A qualitative interview study with carers. Palliat Med. 2018 Sep;32(8):1410-1418. doi: 10.1177/0269216318777656. Epub 2018 Jun 1. PMID 29852808
- [Background] Mehnert A, Lehmann C, Cao P, Koch U. [Assessment of psychosocial distress and resources in oncology--a literature review about screening measures and current developments]. Psychother Psychosom Med Psychol. 2006 Dec;56(12):462-79. doi: 10.1055/s-2006-951828. German. PMID 17160791
- [Background] Zwahlen D, Hagenbuch N, Carley MI, Recklitis CJ, Buchi S. Screening cancer patients' families with the distress thermometer (DT): a validation study. Psychooncology. 2008 Oct;17(10):959-66. doi: 10.1002/pon.1320. PMID 18203146
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Downar J, Goldman R, Pinto R, Englesakis M, Adhikari NK. The "surprise question" for predicting death in seriously ill patients: a systematic review and meta-analysis. CMAJ. 2017 Apr 3;189(13):E484-E493. doi: 10.1503/cmaj.160775. PMID 28385893
- [Derived] Hentschel L, Wellesen A, Krause LC, von Havranek M, Kramer M, Hornemann B, Bornhauser M, Schuler U, Schutte K. Predicting unplanned hospital readmission in palliative outpatients (PRePP) - study protocol of a longitudinal, prospective study to identify informal caregiver-related and structural predictors. BMC Palliat Care. 2022 May 2;21(1):62. doi: 10.1186/s12904-022-00955-y. PMID 35501763